CLINICAL TRIAL: NCT02716805
Title: A Phase 1 Study to Assess Safety and Tolerability of Tremelimumab and Durvalumab, Administered With High Dose Chemotherapy and Autologous Stem Cell Transplant (HDT/ASCT)
Brief Title: Phase 1 Study of Tremelimumab, Durvalumab, High-dose Chemotherapy, + Autologous Stem Cell Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA placed on partial hold due to additional data
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: MedImmune LLC (Industry); Cancer Research Institute, New York City (Other); Multiple Myeloma Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2014-010
Record Dates: First submitted 2016-03-02; First posted 2016-03-23 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma
Keywords: autologous stem cell transplant; HDT/ASCT; CTLA-4; PD-L1; peripheral blood mononuclear cells; PBMC; ASCT
MeSH Terms: conditions — Multiple Myeloma; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — tremelimumab; durvalumab; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Subjects received Prevnar-13 on Day -33 ± 2 days, tremelimumab (75 mg) on Day -31, leukopheresis on ~Day -10, melphalan (200 mg/m^2) on Day -2, ASCT on Day 0, and reinfusion of PBLs and tremelimumab (75 mg) on Day 3. "Late" post-ASCT treatment comprised Prevnar-13 on Days 30 and 60, tremelimumab (75 mg) on Day 100 ± 10 days and Day 128 (Cycles 1 and 2), followed by up to 6 cycles of durvalumab (1500 mg) on Day 1 of Cycles 3 through 8.
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Biological: Prevnar-13; Drug: Melphalan
- Cohort 2 (Experimental): Subjects were to receive Prevnar-13 on Day -33 ± 2 days, tremelimumab (75 mg) on Day -31, leukopheresis on ~Day -10, melphalan (200 mg/m^2) on Day -2, ASCT on Day 0, and reinfusion of PBLs and tremelimumab (75 mg) on Day 3. "Early" post-ASCT treatment comprised Prevnar-13 on Days 30 and 60, tremelimumab (75 mg) on Days 30 through 40 and Day 100 ± 10 days (Cycles 1 and 2), followed by up to 6 cycles of durvalumab (1500 mg) on Day 1 of Cycles 3 through 8.
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Biological: Prevnar-13; Drug: Melphalan
- Cohort 3 (Experimental): Subjects were to receive Prevnar-13 on Day -33 ± 2 days, tremelimumab (75 mg) + durvalumab (1500 mg) on Day -31, leukopheresis on ~Day -10, melphalan (200 mg/m^2) on Day -2, ASCT on Day 0, and reinfusion of PBLs and tremelimumab (75 mg) on Day 3. "Late" post-ASCT treatment comprised Prevnar-13 on Days 30 and 60, tremelimumab (75 mg) + durvalumab (1500 mg) on Day 100 ± 10 days and Day 128 (Cycles 1 and 2), followed by up to 6 cycles of durvalumab (1500 mg) on Day 1 of Cycles 3 through 8.
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Biological: Prevnar-13; Drug: Melphalan
- Cohort 4 (Experimental): Subjects were to receive Prevnar-13 on Day -33 ± 2 days, tremelimumab (75 mg) + durvalumab (1500 mg) on Day -31, leukopheresis on ~Day -10, melphalan (200 mg/m^2) on Day -2, ASCT on Day 0, and reinfusion of PBLs and tremelimumab (75 mg) on Day 3. "Early" post-ASCT treatment comprised Prevnar-13 on Days 30 and 60, tremelimumab (75 mg) + durvalumab (1500 mg) on Days 30 through 40 and Day 100 ± 10 days (Cycles 1 and 2), followed by up to 6 cycles of durvalumab (1500 mg) on Day 1 of Cycles 3 through 8.
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Biological: Prevnar-13; Drug: Melphalan

INTERVENTIONS:
Drug: Tremelimumab — Tremelimumab was administered as an intravenous (IV) infusion over 60 ± 5 minutes at a fixed dose of 75 mg, regardless of weight.
  Other Names: MEDI1123
Drug: Durvalumab — Durvalumab was administered as an IV infusion over 60 ± 5 minutes at a fixed dose of 1500 mg for subjects weighing > 30 kg. If a subject's body weight dropped to ≤ 30 kg on study, the subject was dosed at 600 mg for as long as the body weight remained ≤ 30 kg.
  When applicable, the durvalumab infusion was to start at least 60 minutes after the end of the tremelimumab infusion.
  Other Names: MEDI4736
Biological: Prevnar-13 — Prevnar-13 was administered as an intramuscular injection. The Prevnar-13 dose and the tremelimumab dose were to be separated by a minimum of 48 hours.
Drug: Melphalan — Melphalan was administered as an IV infusion according to institutional standard of care and local prescribing information.

SUMMARY:
This was a Phase 1, open-label, multicenter, study of checkpoint inhibitor therapy (tremelimumab ± durvalumab) prior to and following autologous stem cell transplant (ASCT) and high-dose melphalan in subjects with multiple myeloma who were at a high risk for relapse, were eligible for ASCT, and had available cryopreserved stem cells. Primary study objectives were to determine the safety and tolerability of study treatment. Further objectives were to evaluate the clinical efficacy and biologic activity of the regimen.

DETAILED DESCRIPTION:
Eligible subjects were to be enrolled sequentially into one of 4 treatment cohorts (beginning with Cohort 1) to receive pretreatment with Prevnar-13 on Day -33 ± 2 days, followed by a single dose of tremelimumab (75 mg) administered either alone (Cohorts 1 and 2) or in combination with a single dose of durvalumab (1500 mg; Cohorts 3 and 4) on Day -31 (approximately 21 days prior to steady-state leukopheresis for the collection of autologous peripheral blood lymphocytes [PBLs]). Leukopheresis was performed on Days -10 to -3, followed by high dose therapy (HDT) comprising melphalan (200 mg/m^2) administered intravenously (IV) on Day -2, and ASCT using previously banked hematopoietic stem cells on Day 0. Autologous PBLs were re-infused into subjects on Day +3 following ASCT, with a single dose of tremelimumab (75 mg) administered on the same day. Following HDT/ASCT, treatment was to resume with tremelimumab (75 mg) administered either alone (Cohorts 1 and 2) or in combination with durvalumab (1500 mg; Cohorts 3 and 4) for the first 2 cycles following HDT/ASCT according to the following schedule.

Late post-ASCT treatment:

* Cohort 1: tremelimumab (75 mg) administered alone on Day 100 (±10) and 4 weeks later (Cycles 1 and 2)
* Cohort 3: tremelimumab (75 mg) + durvalumab (1500 mg) administered on Day 100 (±10) and 4 weeks later (Cycles 1 and 2)

Early post-ASCT treatment:

* Cohort 2: tremelimumab (75 mg) administered alone on Days 30 through 40 and Day 100 (±10) (Cycles 1 and 2)
* Cohort 4: tremelimumab (75 mg) + durvalumab (1500 mg) administered on Days 30 through 40 and Day 100 (±10) (Cycles 1 and 2)

For Cycles 3 through 8, durvalumab alone (1500 mg every 4 weeks) was to be administered in all cohorts.

Within each cohort, the second subject did not start treatment until the first subject had completed early engraftment (approximately Day 12 to 18 post-ASCT); therefore, the first subject in each cohort received the first dose of tremelimumab ± durvalumab and was observed for toxicity for approximately 7 weeks prior to enrollment of the second subject.

Protocol-specified dose-limiting toxicities (DLTs) were assessed from the first dose of study treatment up to and including Cycle 2 dosing (Day 128 for Cohorts 1 and 3 or Day 100 for Cohorts 2 and 4). Subjects were not to be treated in a new cohort until all subjects in the previous cohort had completed the DLT evaluation period and ≤ 1 of 6 subjects had experienced DLT.

After enrollment of 6 subjects in Cohort 1, the study was placed on partial clinical hold by the Food and Drug Administration (FDA) due to safety signals observed in other studies investigating pembrolizumab, an anti-programmed cell death-1 (PD-1) antibody, in combination with immunomodulatory agents in subjects with multiple myeloma. As a result, the single subject who was receiving durvalumab during Cycles 3 to 8 discontinued study treatment after Cycle 5; durvalumab was not initiated in the 4 subjects who remained in the study; and no further subjects were enrolled. Upon recommendations from the two Principal Investigators and the study chair, the 4 ongoing subjects, who were in the transplant phase of the study, were permitted to continue post-ASCT tremelimumab treatment after being re-consented under an intermediate expanded access protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed multiple myeloma.
2. Measurable disease either at enrollment, prior to most recent line of salvage therapy, or prior to most recent line of induction therapy. Measurable disease was defined by any of the following:

   * Serum M-spike ≥ 0.5 g/dL
   * Serum free light chain ≥ 10mg/dL
   * Urine monoclonal protein ≥ 200 mg/24 hours
   * Multifocal plasmacytoma
   * ≥ 20% bone marrow plasmacytosis
3. Available CD34+ stem cells (≥ 2 x 10^6/kg).
4. Eligible for autologous stem cell transplantation.
5. Four or less prior lines of systemic therapy for multiple myeloma (induction, first ASCT, consolidation, and maintenance were considered 1 line of therapy unless treatment was modified due to progression of disease as defined by International Myeloma Working Group [IMWG] criteria).
6. Able and willing to provide consent for required bone marrow biopsies.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
8. Anticipated lifespan greater than 3 months.
9. Adequate organ function, as defined below:

   * Total bilirubin within normal ranges unless associated with hepatobiliary metastases or Gilbert syndrome, then total bilirubin ≤ 2 x upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
   * Creatinine ≤ 2.0 mg/dL
   * Carbon monoxide diffusing capacity (DLCO) ≥ 50%
10. Had been informed of other treatment options.
11. Age ≥ 18 years.
12. Able and willing to give valid written informed consent.
13. Body weight > 30 kg.

Exclusion Criteria:

1. Prior exposure to tremelimumab or durvalumab or other anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4), anti-PD-1, anti-programmed cell death ligand-1 (PD-L1) antibodies.
2. History of severe allergic reactions to any unknown allergens or any components of the study drugs.
3. Active or prior autoimmune disease except for autoimmune thyroiditis, vitiligo, or psoriasis not requiring systemic therapy.
4. Prior allogeneic transplantation.
5. Any prior Grade ≥ 3 immune-related adverse event (irAE) or any prior corticosteroid-refractory irAE.
6. Known active or chronic viral hepatitis or history of any type of hepatitis within the last 6 months.
7. History of sarcoidosis syndrome.
8. Active or history of inflammatory bowel disease (colitis, Crohn's), celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea. Active or history of systemic lupus erythematosus or Wegener's granulomatosis.
9. Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, were available.
10. Known immunodeficiency or active human immunodeficiency virus.
11. Other active serious illnesses (e.g., serious infections requiring antibiotics).
12. Prior treatment in any other clinical trial involving another investigational agent within 4 weeks prior to Day -31 of the study; resolution of respective adverse event (AE) to Grade 1 or lower should have occurred.
13. Major surgical procedure (as defined by the Investigator) within 30 days prior to Day -31 or still recovering from prior surgery.
14. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
15. Lack of availability for immunological and clinical follow-up assessments.
16. Women who were breastfeeding or pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]).
17. Female subjects of childbearing potential who were sexually active with a nonsterilized male partner must have used at least one highly effective method of contraception from the time of screening, and must have agreed to continue using such precautions for 90 days after the last dose of durvalumab or for 6 months after the last dose of tremelimumab (whichever was longer). Non-sterilized male partners of a female subject must have used male condoms plus spermicide throughout this period. Cessation of birth control after this point should have been discussed with a responsible physician. Not engaging in sexual activity for the total duration of the trial and the drug washout period was an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method were not acceptable methods of birth control.

    Female subjects should have refrained from breastfeeding throughout the period described above.

    Females of childbearing potential were defined as those who were not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal.

    Females were considered post-menopausal if they had been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements applied:
    * Females < 50 years of age were considered post-menopausal if they had been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they had luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Females ≥ 50 years of age were considered post-menopausal if they had been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

    Women of childbearing potential must have had a negative serum β-HCG pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) conducted during screening and a negative urine β-HCG pregnancy test conducted prior to study drug administration on Day -31. Ongoing serum pregnancy tests were conducted according to the study protocol.

    Nonsterilized male subjects who were sexually active with a female partner of childbearing potential must have used male condoms plus spermicide from screening through 90 days after last dose of durvalumab or through 6 months after the last dose of tremelimumab (whichever was longer). Female partners (of childbearing potential) of a male subject must have used a highly effective method of contraception throughout the period described above. Cessation of birth control after this point should have been discussed with a responsible physician. Not engaging in sexual activity for the total duration of the trial and the drug washout period was an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method were not acceptable methods of contraception.

    Male subjects should have refrained from sperm donation throughout this period. A highly effective method of contraception was defined as one that resulted in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Note that some contraception methods were not considered highly effective (e.g., male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel which was considered highly effective]; and triphasic combined oral contraceptive pills).
18. Any condition that, in the clinical judgment of the treating physician, was likely to prevent the subject from complying with any aspect of the protocol or that may have put the subject at unacceptable risk.
19. Subjects must not have donated blood while on study and for at least 90 days following the last durvalumab treatment or for 6 months following the last tremelimumab treatment, whichever was longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M. Lesokhin, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Research Facility, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: "Late" post-autologous stem cell transplant (ASCT) treatment (tremelimumab alone in Cycles 1-2, durvalumab alone in Cycles 3+)
- Cohort 2: "Early" post-ASCT treatment (tremelimumab alone in Cycles 1-2, durvalumab alone in Cycles 3+)
- Cohort 3: "Late" post-ASCT treatment (tremelimumab + durvalumab in Cycles 1-2, durvalumab alone in Cycles 3+)
- Cohort 4: "Early" post-ASCT treatment (tremelimumab + durvalumab in Cycles 1-2, durvalumab alone in Cycles 3+)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 6 | 0 | 0 | 0
Completed | 4 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Progressive disease | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects.
Groups:
- Cohort 1: "Late" post-ASCT treatment (tremelimumab alone in Cycles 1-2, durvalumab alone in Cycles 3+)
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Eastern Cooperative Oncology Group (ECOG) performance status (PS) [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    0 | 6
    ≥ 1 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from the time of enrollment through the end of the study period. DLTs were assessed from the first dose of study drug through the Cycle 2 administration of tremelimumab ± durvalumab post ASCT. DLTs were defined per protocol as lack of neutrophil/platelet engraftment by Day 30 post ASCT; Grade 5 toxicity (treatment-related death); Grade 4 non-hematological toxicity; Grade 3 non-hematological toxicity (with exclusions); isolated Grade 3 electrolyte abnormalities; or immune-related AEs resulting in discontinuation of treatment.
Time Frame: up to 14 months
Population: All treated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Participants
  Any TEAE | 6
  Maximum grade 2 TEAE | 2
  Maximum grade 4 TEAE | 4
  Immune-related TEAE | 1
  Tremelimumab-related TEAE | 5
  Durvalumab-related TEAE | 1
  Serious TEAE | 1
  TEAE Leading to Treatment Discontinuation | 0
  TEAE Meeting DLT Criteria | 0

2. Secondary Outcome: Number of Subjects With Best Response According to International Myeloma Working Group (IMWG) Consensus Criteria
Description: Response was evaluated by appropriate imaging and myeloma serum/urine tests at the start of Cycle 1 and end of study, with response categorized per IMWG consensus criteria, as follows: stringent complete response (sCR) - CR criteria + normal free light chain (FLC) ratio + no clonal cells in bone marrow; CR - negative immunofixation on serum/urine + no soft tissue plasmacytomas + <5% plasma cells in bone marrow; very good partial response (VGPR) - serum/urine M-protein detectable by immunofixation but not electrophoresis OR ≥90% reduction in serum M-protein + urine <100 mg/24h; PR - ≥50% and ≥90% (or <200 mg/24h) reduction of serum + urine M-protein, respectively; progressive disease - increase of ≥25% serum and/or urine M-component, increase of >10 mg/dL in involved and uninvolved FLC levels, bone marrow plasma cells ≥10%, new or larger lesions, or corrected serum calcium >11.5 mg/dL or 2.65 mmol/L [Rajkumar et al. Blood 2011;117:4691-5; Durie et al. Leukemia 2006;20:1467-73].
Time Frame: Up to 14 months
Population: All subjects who received at least 1 dose of study treatment and underwent at least 1 post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 4
Participants
  sCR | 1
  VGPR | 2
  Progressive disease | 1

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 14 months.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to the indicated study drug; preferred terms were counted only once per subject at the maximum reported grade.
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6)
Acute kidney injury (Renal and urinary disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6)
Nausea (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Blood blister (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 2
Influenza like illness (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Peripheral swelling (General disorders) | 1
Weight decreased (Investigations) | 3
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Thyroxine decreased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Jugular vein occlusion (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Diverticulitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Restlessness (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination due to safety signals in other studies investigating combination regimens comprising similar drugs. Because only 6 subjects were enrolled, no final statistical analysis plan was issued and no formal data analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Main protocol (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT02716805/Prot_SAP_000.pdf
  • Study Protocol: Expanded access protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT02716805/Prot_001.pdf